CLINICAL TRIAL: NCT04351763
Title: Amiodarone or Verapamil in COVID-19 Hospitalized Patients With Symptoms
Acronym: ReCOVery-SIRIO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Eliano Pio Navarese, Prof Eliano P. Navarese, MD, PhD, Nicolaus Copernicus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCU-COVID19
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Amiodarone; Verapamil

STUDY DESIGN:
Intervention Model Description: parallel group, randomized trial
Who Masked: Outcomes Assessor
Masking Description: Clinical events will be validated blindly by an independent clinical event committee (CEC) unaware of the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Amiodarone (Experimental): Amiodarone - administered intravenously
  Bolus of 150 mg is given over a minimum of 10 min, with subsequent continuous infusion of 1 mg/min for 6 h, next continuous infusion of 0.5 mg/min for 18 h, then switch to oral administration.
  Oral administration
  200 to 400 mg/day (adjust dosage based on cardiac response and age) up to discharge.
  Interventions: Drug: Amiodarone
- Verapamil (Experimental): Verapamil - administered intravenously
  Bolus of 0.075-0.15 mg/kg (5-10 mg) over at least 3 minutes, then switch to oral administration.
  Oral administration
  120 to 480 mg/day in divided doses every 6-8 hours (adjust dosage based on cardiac response and age) up to discharge.
  Interventions: Drug: Verapamil
- Usual Care (No Intervention)

INTERVENTIONS:
Drug: Amiodarone — Ion channel blocker
  Arms: Amiodarone
Drug: Verapamil — Ion channel blocker
  Arms: Verapamil

SUMMARY:
There is an urgent need for effective therapies against the novel COVID-19 virus. Studies have shown that amiodarone and verapamil can interfere with coronavirus entry and amplification by blocking ion channels. ReCOVery-SIRIO is a randomized study to investigate amiodarone or verapamil compared with usual care in symptomatic patients hospitalized with confirmed COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients with confirmed COVID-19 infection and symptoms, with an oxygenation index defined as quotient of partial pressure of oxygen in arterial blood (PaO2, in mmHg) and fraction of inspired oxygen (FiO2) > 200.

Exclusion Criteria:

* Acute respiratory distress syndrome (ARDS)
* Contraindications for or known hypersensitivity to amiodarone or calcium channel blockers
* Long QT syndrome
* Prolonged baseline QTc interval (≥450 ms).
* Cardiogenic shock or severe hypotension (SBP< 90 mmHg)
* Severe left ventricle dysfunction (left ventricular ejection fraction ≤35%)
* Severe sinus - node dysfunction with marked sinus bradycardia
* 2nd/3rd degree heart block
* Bradycardia without pacemaker that has caused syncope
* History of severe dysthyroidism
* A-Fib/flutter conducted via accessory pathway (ie,Wolff -Parkinson-White)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | Randomization to day 15
  Time to first occurrence of clinical improvement assessed on a seven category scale ranging from 1 to 7

SECONDARY OUTCOMES:
Clinical improvement | Randomization to day 7 and 28
  Time to first occurrence of clinical improvement assessed on a seven category scale ranging from 1 to 7
Cardiac troponins | 7, 10 and 15 days after randomization
  assessed serially
Mortality | Randomization to day 28
  Individual endpoint
Time to resolution of fever | Randomization to day 28
  Defined as body temperature (≤36.6°C [axilla], or ≤37.2 °C [oral], or ≤37.8°C [rectal]) for at least 48 hours without antipyretics or until discharge, whichever is sooner.
Tachyarrhythmias | Randomization to day 28
  defined as atrial fibrillation, supraventricular or ventricular tachycardia requiring treatment
Time to clinical improvement from admission using the 7-point ordinal scale | Randomization to day 28
  Clinical improvement assessed on a seven category scale ranging from 1 to 7.
Change in NEWS2 score | Randomization to day 7 and 15
  The National Early Warning Score (NEWS2) score. A Higher score is worse.
Duration of hospitalization | Randomization to day 28
  Length of hospitalization in days
PO2/FIO2 | Randomization to day 7 and 15
  oxygenation index defined as quotient of partial pressure of oxygen in arterial blood (PaO2, in mmHg) and fraction of inspired oxygen (FiO2)

CONTACTS AND LOCATIONS:
Locations (1):
- Nicolaus Copernicus University, Bydgoszcz, Poland